CLINICAL TRIAL: NCT01477814
Title: Randomized Clinical Trial to Improve Colon Cancer Screening in Poor Rural Iowa Counties
Brief Title: Interventions to Improve Colon Cancer Screening in Poor Rural Iowa Counties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barcey T. Levy (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor-Investigator, Barcey T. Levy, Professor, IAFP Chair in Rural Medicine, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 200805728
Record Dates: First submitted 2011-11-18; First posted 2011-11-23 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; screening; colonoscopy; fecal immunochemical test; clinical guidelines
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- physician chart reminder (Active Comparator): either a paper or an electronic reminder placed on the subject's medical record to remind the physician to screen for colorectal cancer
  Interventions: Behavioral: Physician chart reminder
- chart reminder, educational mat'ls, FIT (Active Comparator): physician chart reminder plus mailed educational materials, including the Centers for Disease Control CRC Screen for Life, the ACS DVD on CRC screening, a fecal immunochemical test with postage-paid return mailer, a magnet reminding individuals to get screened, and a CRC screening preference sheet where subjects could indicate their preferred CRC test
  Interventions: Behavioral: Physician chart reminder; Behavioral: chart reminder, educational mat'ls, FIT
- CR, ed mat'ls, FIT, phone call (Active Comparator): physician chart reminder (CR) plus mailed educational materials, including the Centers for Disease Control CRC Screen for Life, the ACS DVD on CRC screening, a fecal immunochemical test with postage-paid return mailer, a magnet reminding individuals to get screened, and a CRC screening preference sheet where subjects could indicate their preferred CRC test, and a motivational telephone call designed to elicit barriers and preferences and motivate individuals to complete a CRC screening test.
  Interventions: Behavioral: Physician chart reminder; Behavioral: CR,ed mat'ls, FIT, phone call

INTERVENTIONS:
Behavioral: Physician chart reminder — Subjects randomized to this intervention will have paper or electronic chart reminders placed on their medical records alerting their physicians to the need for colorectal cancer screening
  Other Names: chart reminder
Behavioral: chart reminder, educational mat'ls, FIT — Subjects randomized to this group will have a physician chart reminder, mailed educational packet which includes the CDC Screen for Life materials, a FIT with return envelope, a magnet to remind the subject about CRC screening and a CRC screening preference sheet
  Other Names: chart reminder, mailed education, FIT
  Arms: chart reminder, educational mat'ls, FIT
Behavioral: CR,ed mat'ls, FIT, phone call — Subjects randomized to this group will have a physician chart reminder, mailed educational packet which includes the CDC Screen for Life materials, a FIT with return envelope, a magnet to remind the subject about CRC screening and a CRC screening preference sheet. Subjects will also receive a telephone call from project staff to assess barriers to screening and to encourage CRC screening
  Arms: CR, ed mat'ls, FIT, phone call

SUMMARY:
The goal of the study is to conduct a randomized clinical trial to test several office-based strategies for improving colon cancer screening among individuals who are regular patients at 16 family practice physician offices in the state of Iowa. These offices are members of the Iowa Research Network (IRENE), a rural practice-based research network. The interventions to be tested are increasing in intensity from the usual care provided in the office, to physician chart reminders, mailed educational materials to patients, a fecal immunochemical test with postage-paid return envelope, and a telephone call designed to determine attitudes and barriers to screening, and to motivate subjects to get screened. Our main research questions are: 1)do attitudes toward CRC screening change after providing educational materials about CRC screening? 2)do mailed educational materials and a FIT, with or without a telephone reminder, result in increased rates of CRC testing with the FIT?

DETAILED DESCRIPTION:
Colorectal cancer is the second leading cause of cancer death in the U.S. yet approximately half of eligible adults are not up-to-date with colon cancer screening and the rates of screening are lower among those with lower incomes and who lack insurance. A physician's recommendation for screening has consistently been show to be one of the most powerful predictors of CRC screening. Relatively few studies of CRC screening have been conducted in primary care. Disparities in CRC screening rates are seen in low socioeconomic and rural individuals who often lack resources and access to screening. Most intervention studies have been conducted in managed care settings, community health centers, Veteran's Administration or academic practices. Few studies have looked at interventions in rural medical practices. This research will address screening issues for rural patients and those residing in communities designated as medically underserved. The interventions tested in the study will focus on two key areas: educating the patient about the importance of screening, and reminding the physician about the need to discuss screening during the patient's visit.

The original goal of the study was to enroll 1500 unscreened patients aged 52 to 79 years from 16 family physician practices located in poor, rural Iowa counties. This study will test a combination of patient and physician reminder strategies designed to ensure that the patient is educated about CRC screening and receives a recommendation for CRC screening from their physician. The main outcome is colorectal cancer screening by any of the accepted methods. Rates of screening will be compared across intervention groups. We will also determine how much the interventions cost per person screened.

Patients due for screening within each practice (based on their self-report) (never screened or not up to date with screening) will be randomized to one of four groups that will receive office reminder system strategies of increasing intensity: 1) Usual care, 2) Physician chart reminder alone, 3) Physician chart reminder plus multifaceted mailed patient education, including a postage paid fecal immunochemical test, a reminder magnet, and returnable CRC screening test preference sheet, or 4) Physician chart reminder + multifaceted mailed patient education/FIT/magnet/preference sheet + telephone reminder to encourage screening and address barriers.

Our central hypothesis is that providing offices with one or more CRC screening support systems based on the Chronic Care Model will significantly increase CRC screening rates in comparison with usual care, and that such interventions will be cost-effective and accepted in practice.

ELIGIBILITY:
Inclusion Criteria:

* patients not up-to-date with CRC screening guidelines based on their responses to baseline survey
* patients with a positive personal history of CRC

Exclusion Criteria:

* patients with personal history of CRC or inflammatory bowel disease
* patients with a family history of hereditary conditions that put them at high risk for CRC (familial adenomatous polyposis or hereditary, nonpolyposis CRC)
* inability to read and comprehend the Informed Consent or written survey
* patients who are up-to-date with CRC screening guidelines based on their response to the baseline survey

Ages: 52 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 743 (Actual)
Dates: Start 2008-07; Primary Completion 2010-04-27 (Actual); Study Completion 2015-07-16 (Actual)

PRIMARY OUTCOMES:
colorectal cancer screening | 15 months
  The main outcome measure is the percentage of subjects who complete colorectal cancer screening by any of the accepted methods

SECONDARY OUTCOMES:
cost-effectiveness of various strategies for screening | 15 months
  cost-effectiveness of the various interventions for colorectal cancer screening

CONTACTS AND LOCATIONS:
Overall Officials: Barcey T Levy, PhD, MD, Principal Investigator — University of Iowa
Locations (1):
- Iowa Research Network, University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Written request from an appropriate researcher to the PI

REFERENCES:
- [Background] Levy BT, Xu Y, Daly JM, Ely JW. A randomized controlled trial to improve colon cancer screening in rural family medicine: an Iowa Research Network (IRENE) study. J Am Board Fam Med. 2013 Sep-Oct;26(5):486-97. doi: 10.3122/jabfm.2013.05.130041. PMID 24004700
- [Background] Daly JM, Xu Y, Levy BT. Patients whose physicians recommend colonoscopy and those who follow through. J Prim Care Community Health. 2013 Apr 1;4(2):83-94. doi: 10.1177/2150131912464887. Epub 2012 Nov 4. PMID 23799714
- [Background] Levy BT, Daly JM, Xu Y, Ely JW. Mailed fecal immunochemical tests plus educational materials to improve colon cancer screening rates in Iowa Research Network (IRENE) practices. J Am Board Fam Med. 2012 Jan-Feb;25(1):73-82. doi: 10.3122/jabfm.2012.01.110055. PMID 22218627
- [Background] Ely JW, Levy BT, Daly J, Xu Y. Patient Beliefs About Colon Cancer Screening. J Cancer Educ. 2016 Mar;31(1):39-46. doi: 10.1007/s13187-015-0792-5. PMID 25619196
- [Derived] Daly JM, Xu Y, Ely JW, Levy BT. A randomized colorectal cancer screening intervention trial in the Iowa Research Network (IRENE): study recruitment methods and baseline results. J Am Board Fam Med. 2012 Jan-Feb;25(1):63-72. doi: 10.3122/jabfm.2012.01.110054. PMID 22218626